CLINICAL TRIAL: NCT06270576
Title: Nasal Endotoxin Challenge to Study Mucosal Inflammation in Patients With Asthma
Brief Title: Nasal Inflammation Following Endotoxin Challenge in Patients With Asthma
Acronym: Nasal-LPS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, William Janssen, MD, Section Head of Critical Care, Professor of Medicine, Principle Investigator, National Jewish Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HS3131
Record Dates: First submitted 2024-01-30; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Asthma; Eosinophilic; Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma | interventions — Lipopolysaccharides; Endotoxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Asthma Group (Active Comparator): Subjects diagnosed with one of the three asthma endotypes being studied (T2, T1, or T17).
  Interventions: Drug: Lipopolysaccharides
- Control Group (Active Comparator): Subjects with no diagnosis of asthma or other respiratory disease and are deemed healthy.
  Interventions: Drug: Lipopolysaccharides

INTERVENTIONS:
Drug: Lipopolysaccharides — LPS aka endotoxin is a component of bacterial cell walls and is ubiquitous in the environment. It is found in pet dander, house dust and environmental dusts and has been heavily studied in asthma.
  Other Names: Endotoxin; LPS; Clinical reference center lipopolysaccharide; LPS E. Coli O:113

SUMMARY:
A phase I clinical research study aimed at determining mechanisms that regulate airway mucosal inflammation in asthma endotypes using intranasal administration of endotoxin (lipopolysaccharide from E. coli) in healthy controls and subjects diagnosed with asthma.

DETAILED DESCRIPTION:
Patients with severe asthma can be broadly classified into three endotypes (T2, T1, and T17) based on inflammatory cell and cytokine profiles. Within these endotypes, many patients have high levels of neutrophils in the airways and mucosal epithelium. Our preliminary data suggest that neutrophils in the airways and blood of patients with severe asthma are heterogenous and that subsets exist. The nature of these subsets appears to differ between T2, T1, and T17 asthma endotypes.

In order to advance the field and determine the mechanisms that underpin severe neutrophilic asthma, investigators plan to longitudinally assess transcriptional profiles and functional properties of neutrophil subsets that migrate to the nasal cavity following exposure to a standardized dose of Clinical Reference Center endotoxin (IRB#HS-3131-528, IND 018580).

Investigators will recruit 15 subjects of each asthma endotype (45 total participants with asthma) and 15 healthy controls. LPS will be used to elicit migration of neutrophils into the nasal cavities. Neutrophils will be isolated from the nasal cavities using both nasal lavage and nasal brushes 20 minutes, 1 day and 3 days after endotoxin challenge. Neutrophil biology will be assessed using single-cell RNAseq and ex vivo functional assays.

ELIGIBILITY:
Inclusion Criteria:

* Participants will have asthma diagnosed by a health care provider. Healthy controls are individuals without asthma.
* Written informed consent

Exclusion Criteria:

* Current or recent illness (in the past 4 weeks)
* Recent asthma exacerbation (past 4 weeks)
* History of nasal perforation or nasal surgery
* Nasal polyposis
* Presence or prior history of cardiac or systemic disease
* Bleeding disorder, use of systemic anticoagulants, or antiplatelet therapy
* Immunocompromised state (HIV, immunoglobulin deficiency, systemic immunosuppressants excluding corticosteroids)
* Use of tobacco or marijuana in the past 2 months or greater than a 10 pack-year smoking history
* Currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Neutrophil heterogeneity using single cell RNA sequencing | We anticipate that the study will run over 5 years
  Neutrophil subset composition as determined by single cell RNAseq is compared to endotype groups using a multivariate linear regression framework for compositional data, employing the additive log ratio transformation. Models will include indicator variables for whether a sample is T1 high, T2 high, T17 high or non-asthmatic and will control for age, sex, and smoking status. AM subset gene expression matrices from scRNAseq will be compared between endotypes using the pseudo bulk approach to account for clustering of cells within subjects. To identify global gene expression programs underlying each endotype, bulk RNAseq gene expression data will be normalized using DESeq2's variance stabilizing transformation and similarly compared between endotypes using linear regression models. A Benjamini-Hochberg adjustment will be used to control the false discovery rate.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No